CLINICAL TRIAL: NCT06904482
Title: Co-Transplant of an Unmodified Haplo-Identical Graft With Cord Blood
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE9Z24
Record Dates: First submitted 2025-03-31; First posted 2025-04-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: aGVHD; Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndromes
Keywords: Unmodified Haplo-Identical Graft with Cord Blood; post-transplant cyclophosphamide aGVHD prophylaxis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Haplo-Identical / Cord Blood Transplant (Experimental)
  Interventions: Biological: Haplo-Identical / Cord Blood Transplant

INTERVENTIONS:
Biological: Haplo-Identical / Cord Blood Transplant — Cord Blood Unit Selection Cord Blood Unit Selection should be consistent with published guidelines5 with the understanding that the goal cell dose is 1x105 CD34 cells/kg in this protocol. ABO matching and donor specific antibodies should be taken into account in the selection of the CB unit.
  Haplo-Donor Selection Haplo-identical siblings and younger male donors are preferred. ABO matching, CMV compatibility, and donor specific antibodies should be taken into account in the selection of the donor.

SUMMARY:
The purpose of this study is to see if see if adding the specific combination of donors can result in acceptable levels of survival without evidence of disease.

DETAILED DESCRIPTION:
Cord blood (CB) and haplo-identical grafts are valuable alternative graft sources for patients with hematologic malignancies in need of allogeneic transplantation who lack human leukocyte antigen (HLA)-matched adult donors. In Black, Asian, Hispanic populations, the chance of finding a HLA matched donor is 23%, 41%, and 46%, respectively. These graft sources allow for greater HLA difference between donor and recipient, and increase the availability of donors, and therefore transplant, to these populations. Comparative retrospective analyses demonstrate similar results when compared to haplo/cord transplants. In this variant of the standard haplo/cord transplant, investigators will utilize post-transplant cyclophosphamide aGVHD prophylaxis after infusion of the haplo-identical graft and then infuse the CB graft after completion of post-transplant cyclophosphamide. Our hypothesis is that the combination of these two graft sources in which the haplo-identical graft is unmanipulated and the CB graft is infused after post-transplant cyclophosphamide, will be safe and result in effective disease eradication as measured by progression free survival in high risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with the following hematologic malignancies:

   * Acute myelogenous leukemia (AML): High-risk AML including:

     * Antecedent hematological disease (e.g., myelodysplasia (MDS))
     * Treatment-related
     * Complete Remission (CR1) with poor or intermediate-risk cytogenetics or molecular markers (e.g. Flt 3 mutation, 11q23, del 5, del 7, TP53 mutations, complex cytogenetics)
     * Participant must be in CR1, CR2, CR3 or CRi
   * Acute lymphoblastic leukemia (ALL)

   High-risk CR1 including:
   * Poor-risk cytogenetics (e.g., t(9;22)or 11q23 rearrangements)
   * Presence of minimal disease by flow cytometry or PCR or Clonoseq after 2 or more cycles of chemotherapy
   * No CR within 4 weeks of initial treatment Participant must be in CR1, CR2, CR3, or CRi

     * Myelodysplastic syndromes (MDS), Intermediate, High or Very High Risk by the revised international prognostic scoring system (IPSS-R) or treatment related MDS.
2. Age > 18 years
3. Participants without a suitable HLA-matched related or unrelated donor
4. Participant with the following suitable grafts:

   * A 4-8/8 HLA high resolution matched CB unit with a cell dose of 1.0x105 CD34 cells/kg.
   * A haplo-identical donor with a goal cell dose of > 4.0x106 CD34cells/kg (minimum 2 x106 CD34/kg)
5. Concurrent Therapy for Extramedullary Leukemia or CNS Lymphoma: Concurrent therapy or prophylaxis for testicular leukemia, CNS leukemia including standard intrathecal chemotherapy and/or radiation therapy will be allowed as clinically indicated. Such treatment may continue until the planned course is completed. Participants must be in CNS remission at the time of protocol enrollment if there is a history of CNS involvement. Maintenance therapy after transplant is allowed.
6. Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Participants with inadequate Organ Function as defined by:

   * Creatinine clearance < 40ml/min (Cockcroft-Gault)
   * Bilirubin > 2X institutional upper limit of normal unless Gilbert syndrome
   * AST (SGOT) > 3X institutional upper limit of normal
   * ALT (SGPT) > 3X institutional upper limit of normal
   * Pulmonary function: DLCOc < 60%
   * Cardiac: left ventricular ejection fraction < 40%
   * ECOG <2
2. Participants with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Pregnant or breastfeeding women are excluded from this study because chemotherapy involved with RIC have the significant potential for teratogenic or abortifacient effects.
4. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
5. Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.
6. Prior autologous stem cell transplant or CAR-T within the preceding 6 months or prior allogeneic transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2027-02-24 (Estimated); Study Completion 2030-02-25 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) at 6 months after transplant | 6 months after transplant
  Kaplan-Meier method will be used to estimate the PFS

SECONDARY OUTCOMES:
Progression free survival at 1 year after transplant | 1 year after transplant
  Kaplan-Meier method will be used to estimate the PFS
Progression free survival at 2 years after transplant | 2 years after transplant
  Kaplan-Meier method will be used to estimate the PFS
Progression free survival at 3 years after transplant | 3 years after transplant
  Kaplan-Meier method will be used to estimate the PFS
Non-relapse mortality at 1 year after transplant | 1 year after transplant
Non-relapse mortality at 2 years after transplant | 2 years after transplant
Non-relapse mortality at 3 years after transplant | 3 years after transplant
Overall survival(OS) at 1 year after transplant | 1 year after transplant
  Kaplan-Meier method will be used to estimate the OS
Overall survival at 2 years after transplant | 2 years after transplant
  Kaplan-Meier method will be used to estimate the OS
Overall survival at 3 years after transplant | 3 years after transplant
  Kaplan-Meier method will be used to estimate the OS
Graft versus host disease relapse free survival at 1 year after transplant | 1 year after transplant
Graft versus host disease relapse free survival at 2 years after transplant | 2 years after transplant
Graft versus host disease relapse free survival at 3 years after transplant | 3 years after transplant
Relapse at 1 year after transplant. | 1 year after transplant.
Relapse at 2 years after transplant. | 2 years after transplant.
Relapse at 3 years after transplant. | 3 years after transplant.
Rate of grade III-IV Acute Graft Versus Host Disease (aGVHD) at 30 days after transplant | 30 days after transplant
Rate of grade III-IV aGVHD at 100 days after transplant | 100 days after transplant
Rate of grade III-IV aGVHD at 6 months after transplant | 6 months after transplant
Rate of grade III-IV aGVHD at 1 year after transplant | 1 year after transplant
Rate of grade III-IV aGVHD at 2 years after transplant | 2 years after transplant
Rate of grade III-IV aGVHD at 3 years after transplant | 3 years after transplant
Rate of grade II-IV aGVHD at 30 days after transplant | 30 days after transplant
Rate of grade II-IV aGVHD at 100 days after transplant | 100 days after transplant
Rate of grade II-IV aGVHD at 6 months after transplant | 6 months after transplant
Rate of grade II-IV aGVHD at 1 year after transplant | 1 year after transplant
Rate of grade II-IV aGVHD at 2 years after transplant | 2 years after transplant
Rate of grade II-IV aGVHD at 3 years after transplant | 3 years after transplant
Rate of severe Chronic Graft Versus Host Disease (cGVHD) at 100 days after transplant. | 100 days after transplant
Rate of severe cGVHD at 6 months after transplant. | 6 months after transplant
Rate of severe cGVHD at 1 year after transplant. | 1 year after transplant
Rate of severe cGVHD at 2 years after transplant. | 2 years after transplant
Rate of severe cGVHD at 3 years after transplant. | 3 years after transplant
Rate of moderate cGVHD at 100 days after transplant | 100 days after transplant
Rate of moderate cGVHD at 6 months after transplant | 6 months after transplant
Rate of moderate cGVHD at 1 year after transplant | 1 year after transplant
Rate of moderate cGVHD at 2 years after transplant | 2 years after transplant
Rate of moderate cGVHD at 3 years after transplant | 3 years after transplant
Rate of mild cGVHD at 100 days after transplant | 100 days after transplant
Rate of mild cGVHD at 6 months after transplant | 6 months after transplant
Rate of mild cGVHD at 1 year after transplant | 1 year after transplant
Rate of mild cGVHD at 2 years after transplant | 2 years after transplant
Rate of mild cGVHD at 3 years after transplant | 3 years after transplant
Rate of serious infections at 1 year after transplant | 1 year after transplant
Time to neutrophil engraftment. | 60 days post treatment
  Neutrophil engraftment will be calculated as the days from transplant where the absolute neutrophil count (ANC) reaches >500cells/ul x 3 days.
Time to platelet engraftment. | 60 days post treatment
  Platelet engraftment will be calculated as the days from transplant where the platelet count reaches 20,000 platelets /ul without the need of transfusion of platelets for 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals Cleveland Medical Center
Locations (1):
- Case Comprehensive Cancer Center, University Hospitals Cleveland Medical Center Seidman Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed participant data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan.